CLINICAL TRIAL: NCT04417478
Title: Effect of Periodontal Debridement on Leptin Levels in Patients With Class I and II Obesity With Periodontitis
Brief Title: Effect of Periodontal Debridement on Leptin Levels in Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Mariely Navarrete, Associate Professor, Faculty of Dentistry Andres Bello University, Viña del Mar campus, Universidad Nacional Andres Bello
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Periodontitis; Obesity
Keywords: Obesity; Periodontal debridement; Periodontitis; Leptin; Body mass index
MeSH Terms: conditions — Periodontitis; Obesity | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: A double-blind, controlled, clinical trial was conducted. The sampling method was probabilistic stratified and the sample size 27 subjects in total, divided in 3 groups of: 9 normal weight patients, 9 class I Obesity patients and 9 class II Obesity patients and history of moderate to severe periodontitis, who met the inclusion and exclusion criteria and signed an informed consent. All patients received SRP and clinical monitoring at baseline and 3 months post-therapy by the same examiner.Serum levels of leptin were evaluated by enzyme-linked immunosorbent assay at baseline and 3 months post SRP by one trained examiner.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal weight (Active Comparator): Patients with Periodontitis and normal weight, that is BMI fluctuates between 18,50 y 24,99 kg/m2.
  Interventions: Other: Scaling and root planning
- class I Obesity (Experimental): Patients with Periodontitis and class I Obesity, that is BMI fluctuates between 30,00 a 34,99 kg/m2.
  Interventions: Other: Scaling and root planning
- class II Obesity (Experimental): Patients with Periodontitis and class II Obesity, that is BMI fluctuates between 35,00 y 39,99 kg/m2.
  Interventions: Other: Scaling and root planning

INTERVENTIONS:
Other: Scaling and root planning — Periodontal debridement was performed in all patients.

SUMMARY:
The main purpose of the study is to quantify of Leptin hormone in patients with normal weight, class I obesity, class II obesity and periodontitis, before and after scaling and root planning (SRP) and correlate the Body mass index (BMI) with Leptin levels.

A double-blind, controlled, clinical trial was conducted. The sampling method was probabilistic stratified and the sample size 27 subjects in total, divided in 3 groups of: 9 normal weight patients, 9 class I Obesity patients and 9 class II Obesity patients and history of Generalized Periodontitis Stage II,III or IV, Grade B or C, who met the inclusion and exclusion criteria and signed an informed consent.

All patients received SRP and clinical monitoring at baseline and 3 months post-therapy by the same examiner.Probing depth (PD), Clinical Attachment Level (CAL), Biofilm Index (BI) and Bleeding on Probing (BoP), Tooth Mobility and Suppuration were evaluated as clinical variables. Serum levels of leptin were evaluated by enzyme-linked immunosorbent assay (ELISA) at baseline and 3 months post SRP.

DETAILED DESCRIPTION:
Definition of the sample: 30 patients were recruited from the Diagnosis Unit of Andres Bello University Faculty of Dentistry (DUFD), campus Viña del Mar, with the diagnosis of Generalized Periodontitis Stage II, III or IV, grade B or C who were catalogued as normal weight, class I obesity and class II obesity who also fulfill the inclusion and exclusion criteria. Once the patients accepted the invitation to participate in the Investigative Project, they were given all the details and were requested to sign the Informed Consent form.

Sample Size Calculation:The minimum sample size necessary to validate the investigation is based on the study and results explained by Gonçalves, et al (2015), based on the variance of the differences of BMI of each classification. Considering the former data and using a significance level of 1%, a statistical power of 90% and an estimation error of 1, it was estimated a minimum of 12 patients for each group of normal weight, class I obesity and class II obesity. With the purpose of making a noticeable distinction between groups (class I and class II obesity) and without affecting the results of this study, there were considered 10 patients for each group of study.

Protocol and clinical exam: From the 30 initial patients at the beginning of the study, 27 was the number of patients who finally participated in it, as a result of 1 loss of tracing and 2 patients who interrupted their treatment. Two experimental groups were formed considering class I and class II obesity patients. The third group had control purposes and was composed by normal weight patients.

Presence or not of Obesity was determined by BMI, an indicator according to World Health Organization (WHO) which classifies adult population in several categories of weight using height and weight data. This information was measured and registered by only one examiner within the study. No compliance problems were noted and all patients followed the protocol of the study. None subjects reported specific adverse effects.

Type and design of study Randomized Clinical Trial. Sampling method: Probabilistic Stratified. Sample size: 27 subjects in total, divided in 3 groups of: 9 normal weight patients, 9 class I Obesity patients and 9 class II Obesity patients.

Standardization and calibration: In order to execute a properly standardized process, only instruments and supplies of the same commercial brand were used: periodontal diagnosis was always performed in a determined dental chair at the Dental Clinic of DUFD, under the same lighting system using a North Carolina Periodontal Probe (Hu-Friedy® Manufacturing Inc., Chicago,Illinois,USA). Only one examiner (FP) performed diagnosis and anthropometric measurements; these last ones were measured in a weight scale and measuring tape at the Dental Clinic of DUFD.

An inter-examiner calibration was necessary for diagnostic purposes and periodontal charting. This was performed between the only one examiner (FP) calibrated by the principal investigator (MN) according to a record set of calibration, which evaluated 2 sites in 4 teeth in a specific individual. This data was analysed according to Lin's Concordance Correlation Coefficient.

Anthropometric Measurements: An only one examiner inquired all measures of weight (Kg) and height (cm). BMI was calculated dividing weight by the height square. Patients were catalogued in a normal weight range when their BMI fluctuated between 18,50 y 24,99 kg/m2, Class I Obesity with a BMI between 30,00 a 34,99 kg/m2 and Class II Obesity with a BMI between 35,00 y 39,99 kg/m2, according to WHO.

Periodontal debridement: Patients were instructed according to Modified Bass Brushing Technique and were provided with the necessary items to do it properly (Dentaid® toothbrush, toothpaste and interdental brush). An exclusive examiner (IP) performed supragingival and subgingival debridement consistent in biofilm and dental calculus removal using an ultrasonic scaler (DTE®, Guilin Woodpecker Medical Instrument Co., Ltd., Guilin, Guangxi, P.R. China), followed by root scaling and planing in sites with Probing Depth ≥ 5mm and Clinical Attachment Level ≥ 4mm, using Gracey curettes (Hu-Friedy® Manufacturing Inc., Chicago, Illinois, USA). This treatment was performed to all patients taking 1-2 hours of work within 2- 4 maximum sessions. The procedures were performed under local anesthesia. Patients were called to a check-up at 3 months after treatment.

Clinical Evaluation : Patients went through a clinical evaluation at the beginning of treatment and after 3 months since therapy. The periodontal chart was completed using a North Carolina Periodontal Probe (Hu-Friedy® Manufacturing Inc., Chicago, Illinois, USA) measuring PD, CAL, presence of biofilm, bleeding on probing, suppuration and mobility.

Serum samples: All patients went through a blood sample collection consisting in the extraction of 4 millilitres of peripheral venous blood of the antecubital fascia of the arm with a 20-gauge needle and kept on stored in 6 millilitres serum Becton Dickinson (BD)Vacutainer® tubes. An hour after this process, the blood sample was centrifuged at 4000 revolutions per minute (rpm)for 10 minutes separating this way the rest of the components of the blood, which were distributed in aliquots and stored in -80 degree Celsius (ºC) for further analysis.

ELISA: One trained examiner (IP) analysed the serum samples by using the Leptin ELISA Kit (Thermo Fisher Scientific®., Massachusetts, USA). The trials were done according to manufacturer's instructions. This ELISA Kit is based on the "sandwich" technique for ELISA, it is to say, antibodies against a specific antigen coating the walls of the recipients of the ELISA kit. Since this kit works by immunoadsorption, the colour intensity of the product was directly proportional to the antigen concentration present in the sample. The optical density of the plate reader was adjusted to 450 mm. The results were measured as the concentration in milliliters of serum (pg/mL).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years.
* Patients classified by the American Society of Anesthesiologists (ASA) as ASA I or ASA II that are compatible with local anaesthesia procedures; - Present at least 10 natural teeth, excluding semi-erupted third molars.
* Present at least 6 sites with a probing depth (PD) ≥ 5mm and clinical attachment loss (CAL) ≥ 4mm.
* BMI between 18,50 - 39,99 kg/m2.

Exclusion Criteria:

* Patients with hemostasis disorders.
* Patients who use any medication associated with gingival disorders such as: Anticonvulsants (Phenytoin), Calcium channel blockers (Nifedipine), Immunosuppressive drugs (Cyclosporins).
* Patients with systemic diseases that affect the immunoinflammatory response.
* Patients under treatment with drugs such as: warfarin, digoxin and acetylsalicylic acid.
* Previous history of allergy to local anesthetics.
* Patients who suffer from systemic conditions that can affect the progression of periodontitis and/or the gain or loss of weight, for example:

Diabetes Mellitus, immunological disorders, hypothyroidism,etc.

* Patients who are under weight loss treatment (pharmacological, diet, exercise,etc).
* Patients presenting orthodontic appliances.
* Patients who have received antibiotic or periodontal treatment in the last 3 months.
* Pregnancy.
* Carriers of valvular prostheses or failures in heart valves, with endocarditis risk.
* Patients who are psychically and intellectually incapacitated to participate, according to the Chilean law number 20,584, title II, paragraph 8, article 28.
* Heavy smoking patients, which is smoking more than 10 cigarettes per day.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Difference in serum levels of leptin at baseline and 3 month after SRP, in periodontal patients with normal weight, class I obesity and class II obesity. | Baseline and 3 month
  Before and 3 month after performing SRP, serum levels of leptin was measured. All patients went through a blood sample collection consisting in the extraction of 4 milliliters of peripheral venous blood of the antecubital fossa of the arm with a 20-gauge needle and kept on stored in 6 milliliters serum Becton Dickinson (BD) Vacutainer® tubes. An hour after this process, the blood sample was centrifuged at 4000 rpm for 10 minutes separating this way the rest of the components of the blood, which were distributed in aliquots and stored in -80 degree Celsius (ºC) for further analysis. Later, the serum samples were analysed by using the Leptin ELISA Kit (Thermo Fisher Scientific®., Massachusetts, USA).
  The results were measured as the concentration in millilitres of serum leptin (pg/ml).The student t test and ANOVA were applied to observe if there were significant differences between treatment groups.

SECONDARY OUTCOMES:
Relation between serum levels of leptin and BMI of the periodontal patients, at baseline and 3 months after SRP. | Baseline and 3 month
  Before and 3 months after performing SRP, serum levels of leptin were measured in the same way as described for the primary results.
  BMI was calculated dividing weight by the height square. Patients were catalogued in a normal weight range when their BMI fluctuated between 18,50 y 24,99 kg/m2, Class I Obesity with a BMI between 30,00 a 34,99 kg/m2 and Class II Obesity with a BMI between 35,00 y 39,99 kg/m2, according to WHO. It was performed a correlation analysis using Kendall Tau test.
Number of sites with PD 1-3, 4-6 and ≥ 7mm and CAL ≥ 4 mm in periodontal patients obese and non obese, at baseline and 3 months after SRP. | Baseline and 3 month.
  PD corresponds to the distance in millimetres from the gingival margin (MG) to the inserted probe´s tip of the most apical portion of the periodontal pocket and CAL corresponds to the distance measured in millimetres from the cementum enamel junction to the tip of the probe inserted to the most apical portion of the periodontal pocket.Both were obtained by measuring with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, Illinois, USA), in a position parallel to the vertical axis of the tooth, with a pressure no greater than 0.25 Newtons (N), in a circular direction over the entire surface of each tooth, registering the 6 deepest sites per tooth (mesiobuccal, buccal, distobuccal,distolingual, lingual and mesiolingual). Subsequently, those sites were counted and the student t test was applied to observe if there were significant differences between both treatment groups.
Difference in the Biofilm Index (BI) in periodontal patients obese and non obese, at baseline and 3 months after SRP. | Baseline and 3 month.
  BI is percentage of dental surfaces with staining, through the use of biofilm developers. To obtain the index, a curaprox developer tablet was dissolved in a plastic cup with water and with a cotton ball this solution was applied on all of the tooth surfaces, recording only those that were stained. The calculation was made by dividing the surfaces that stained by the total surfaces, which corresponds to the number of teeth present multiplied by 4, and multiplying this value by 100. Subsequently, student t test was applied to observe if there were significant differences between treatment groups.
Difference in Bleeding on Probing (BoP) index and Suppuration, in periodontal patients obese and non obese, at baseline and 3 months after SRP. | Baseline and 3 month.
  BoP is the percentage of sites that bleed when probing. Suppuration corresponds to the exit of purulent exudate by the crevice.
  Both were recorded during PD measurement with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, Illinois, USA) and was considered positive if it occurs 20 seconds after probing. The calculation was made by dividing the sites that bled or has suppuration by the total sites, which corresponds to the number of teeth present multiplied by 6, and multiplying this value by 100. Subsequently, student t test was applied to observe if there were significant differences between treatment groups.

OTHER OUTCOMES:
Presence of Tooth Mobility grade I, II or III in periodontal patients obese and non obese, at baseline and 3 months after SRP. | Baseline and 3 month.
  Tooth Mobility it is measured clinically by applying pressure with the ends of 2 metal instruments and trying to rock a tooth gently in a bucco-lingual or palatine direction.
  Grade 1: Perceptible mobility <1mm in bucco- lingual or palatine direction. Grade 2: >1mm but < 2mm. Grade 3: >2mm or depressibility in the socket.

CONTACTS AND LOCATIONS:
Overall Officials: Mariely Navarrete Riffo, MSc, Principal Investigator — Universidad Nacional Andres Bello
Locations (1):
- Universidad Nacional Andres Bello, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Jain H, Mulay S. Relationship between periodontitis and systemic diseases: leptin, a new biomarker? Indian J Dent Res. 2014 Sep-Oct;25(5):657-61. doi: 10.4103/0970-9290.147118. PMID 25511069
- [Background] Papageorgiou SN, Reichert C, Jager A, Deschner J. Effect of overweight/obesity on response to periodontal treatment: systematic review and a meta-analysis. J Clin Periodontol. 2015 Mar;42(3):247-61. doi: 10.1111/jcpe.12365. Epub 2015 Feb 20. PMID 25580635
- [Result] Goncalves TE, Zimmermann GS, Figueiredo LC, Souza Mde C, da Cruz DF, Bastos MF, da Silva HD, Duarte PM. Local and serum levels of adipokines in patients with obesity after periodontal therapy: one-year follow-up. J Clin Periodontol. 2015 May;42(5):431-9. doi: 10.1111/jcpe.12396. Epub 2015 Apr 30. PMID 25858047